CLINICAL TRIAL: NCT01330316
Title: A Phase III, Open-label Study of Once Daily BI 201335 240 mg for 24 Weeks in Combination With Pegylated interferon-a (PegIFN) and Ribavirin (RBV) in Patients With Genotype 1 Chronic Hepatitis C Infection Who Failed a Prior PegIFN / RBV Treatment
Brief Title: A Rollover Study of BI 201335 in Combination With Pegylated Interferon-alpha and Ribavirin in Treatment-experienced Genotype 1 Hepatitis C Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1220.48; 2011-000141-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2011-04-05; First posted 2011-04-06 (Estimated); Results first posted 2015-07-31 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — faldaprevir

ARMS (1):
- BI 201335 for 24 weeks (Experimental): BI 201335 once daily dose for 24 weeks in combination with PegIFN/RBV for 24 or 48 weeks
  Interventions: Drug: BI 201335; Drug: PegIFN/RBV

INTERVENTIONS:
Drug: BI 201335 — BI 201335 for 24 weeks
Drug: PegIFN/RBV — PegIFN/RBV for 48 weeks

SUMMARY:
The objective of this trial is to collect evidence for the safety and efficacy of 24 weeks of treatment with BI 201335 240 mg in combination with 24 or 48 weeks of Pegylated Interferon (PegIFN) and ribavirin (RBV) in treatment experienced patients who have been withdrawn from PegIFN and RBV treatment due to lack of efficacy in the 1220.7, 1220.30 and 1220.47 trials.

ELIGIBILITY:
Inclusion criteria:

Chronic hepatitis C infection of GT-1 in patients who failed prior treatment with PegIFN and RBV in the 1220.7, 1220.30 and 1220.47 trials of the BI 201335 Phase III program.

1. Patients from trials 1220.7, 1220.30 and 1220.47 of BI 201335 who have failed treatment with PegIFN/RBV in the placebo groups due to protocol-defined criteria of treatment failure (i.e. either non-response on treatment or relapse after end of treatment [EOT]).
2. Patients must have received at least 4 weeks of assigned trial medication and been compliant with all study procedures.
3. Female patients:

   * with documented hysterectomy,
   * who have had both ovaries removed,
   * with documented tubal ligation,
   * who are post-menopausal with last menstrual period at least 12 months prior to screening, or
   * of childbearing potential with a negative serum pregnancy test at screening and Day 1, that, if sexually active, agree to use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of RBV in addition to the consistent and correct use of a condom. Patients must agree not to breast-feed at any time from the date of screening until 7 months after the last dose of RBV.

   Medically accepted methods of contraception for females in this trial are ethinyl estradiol-containing contraceptives, diaphragm with spermicide substance, intra-uterine device and cervical cap.

   or

   Male patients:
   * who are documented to be sterile, or
   * who are without pregnant female partner(s) and consistently and correctly use a condom while their female partner(s) (if of child-bearing potential) agree to use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin. It is in the responsibility of the male patient to ensure that his partner(s) is not pregnant prior to screening into the study or becomes pregnant during the treatment and the observation phase. Female partners of childbearing potential must perform monthly pregnancy tests from the date of screening until 7 months after the last dose of ribavirin (tests will be provided by the sponsor).
4. Signed informed consent form prior to trial participation.

Exclusion criteria:

1. Evidence of acute or chronic liver disease due to causes other than chronic HCV infection. Incidental steatosis diagnosed by biopsy is not an exclusion criteria.
2. HIV co-infection
3. Hepatitis B virus (HBV) infection based on presence of HBs-Ag
4. Active malignancy, or history of malignancy within the last 5 years prior to screening (with an exception of appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix)
5. Active or, history of alcohol or illicit drug abuse other than cannabis within the past 12 months
6. A condition that is defined as one which in the opinion of investigator may put the patient at risk because of participation in this study, may influence the results of this study, or limit the patients ability to participate in this study
7. Usage of any investigational drugs within 30 days prior to screening, or planned usage of an investigational drug during the course of this study.
8. Received concomitant systemic antiviral, hematopoietic growth factor, or immunomodulatory treatment within 30 days prior to screening. Patients being treated with oral antivirals such as acyclovir, famciclovir or valacyclovir for recurrent herpes simplex infection; or with oseltamivir or zanamivir for influenza A infection, may be screened.
9. Received silymarin (milk thistle), glycyrrhizin, or Sho-saiko-to (SST) within 28 days prior to enrolment and throughout the treatment phase of this trial.
10. Known hypersensitivity to any ingredient of the study drugs.
11. Alpha fetoprotein value > 100 ng/mL at screening; if > 20 ng/mL and = 100 ng/mL, patients may be included if there is no evidence of liver cancer in an appropriate imaging study (e.g., ultrasound, CT scan, or MRI) within last 6 months prior to randomization (Visit 2).

Other exclusion criteria related to pegylated interferon and/or ribavirin restrictions are not listed here.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2011-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (87):
- United States (20):
  - 1220.48.0004 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1220.48.0091 Boehringer Ingelheim Investigational Site, North Little Rock, Arkansas
  - 1220.48.0011 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1220.48.0018 Boehringer Ingelheim Investigational Site, Oceanside, California
  - 1220.48.0078 Boehringer Ingelheim Investigational Site, Fort Lauderdale, Florida
  - 1220.48.0095 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 1220.48.0039 Boehringer Ingelheim Investigational Site, Columbus, Georgia
  - 1220.48.0013 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1220.48.0087 Boehringer Ingelheim Investigational Site, Baton Rouge, Louisiana
  - 1220.48.0027 Boehringer Ingelheim Investigational Site, Framingham, Massachusetts
  - 1220.48.0065 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1220.48.0023 Boehringer Ingelheim Investigational Site, Tupelo, Mississippi
  - 1220.48.0066 Boehringer Ingelheim Investigational Site, Neptune City, New Jersey
  - 1220.48.0012 Boehringer Ingelheim Investigational Site, New York, New York
  - 1220.48.0058 Boehringer Ingelheim Investigational Site, Portland, Oregon
  - 1220.48.0063 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1220.48.0029 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1220.48.0017 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1220.48.0071 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1220.48.0081 Boehringer Ingelheim Investigational Site, Forth Worth, Texas
- Austria (2):
  - 1220.48.4301 Boehringer Ingelheim Investigational Site, Vienna
  - 1220.48.4302 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (3):
  - 1220.48.3201 Boehringer Ingelheim Investigational Site, Brussels
  - 1220.48.3204 Boehringer Ingelheim Investigational Site, Edegem
  - 1220.48.3203 Boehringer Ingelheim Investigational Site, Liège
- Canada (7):
  - 1220.48.1012 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1220.48.1003 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.48.1016 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1220.48.1007 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1220.48.1009 Boehringer Ingelheim Investigational Site, Winnipeg, Manitoba
  - 1220.48.1005 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1220.48.1006 Boehringer Ingelheim Investigational Site, Toronto, Ontario
- France (7):
  - 1220.48.3301 Boehringer Ingelheim Investigational Site, Clichy
  - 1220.48.3311 Boehringer Ingelheim Investigational Site, Lille
  - 1220.48.3303 Boehringer Ingelheim Investigational Site, Marseille
  - 1220.48.3304 Boehringer Ingelheim Investigational Site, Montpellier
  - 1220.48.3305 Boehringer Ingelheim Investigational Site, Nice
  - 1220.48.3316 Boehringer Ingelheim Investigational Site, Pessac
  - 1220.48.3312 Boehringer Ingelheim Investigational Site, Saint-Laurent-du-Var
- Germany (9):
  - 1220.48.4902 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.48.4904 Boehringer Ingelheim Investigational Site, Berlin
  - 1220.48.4913 Boehringer Ingelheim Investigational Site, Dortmund
  - 1220.48.4906 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1220.48.4901 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1220.48.4908 Boehringer Ingelheim Investigational Site, Hamburg
  - 1220.48.4914 Boehringer Ingelheim Investigational Site, Kiel
  - 1220.48.4911 Boehringer Ingelheim Investigational Site, Mainz
  - 1220.48.4905 Boehringer Ingelheim Investigational Site, München
- Japan (8):
  - 1220.48.8106 Boehringer Ingelheim Investigational Site, Chiba, Chiba
  - 1220.48.8117 Boehringer Ingelheim Investigational Site, Kita-gun, Kagawa
  - 1220.48.8116 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 1220.48.8118 Boehringer Ingelheim Investigational Site, Kurume, Fukuoka
  - 1220.48.8113 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1220.48.8114 Boehringer Ingelheim Investigational Site, Nishinomiya, Hyogo
  - 1220.48.8119 Boehringer Ingelheim Investigational Site, Omura, Nagasaki
  - 1220.48.8121 Boehringer Ingelheim Investigational Site, Osaka, Osaka
- Portugal (4):
  - 1220.48.3503 Boehringer Ingelheim Investigational Site, Aveiro
  - 1220.48.3509 Boehringer Ingelheim Investigational Site, Barreiro
  - 1220.48.3501 Boehringer Ingelheim Investigational Site, Lisbon
  - 1220.48.3502 Boehringer Ingelheim Investigational Site, Porto
- 1220.48.4002 Boehringer Ingelheim Investigational Site, Bucharest, Romania
- Russia (2):
  - 1220.48.7001 Boehringer Ingelheim Investigational Site, Moscow
  - 1220.48.7004 Boehringer Ingelheim Investigational Site, Moscow
- South Korea (5):
  - 1220.48.8204 Boehringer Ingelheim Investigational Site, Pusan
  - 1220.48.8205 Boehringer Ingelheim Investigational Site, Pusan
  - 1220.48.8206 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.48.8207 Boehringer Ingelheim Investigational Site, Seoul
  - 1220.48.8201 Boehringer Ingelheim Investigational Site, Yangsan
- Spain (10):
  - 1220.48.3406 Boehringer Ingelheim Investigational Site, A Coruña
  - 1220.48.3402 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.48.3404 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.48.3411 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.48.3412 Boehringer Ingelheim Investigational Site, Barcelona
  - 1220.48.3405 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.48.3409 Boehringer Ingelheim Investigational Site, Madrid
  - 1220.48.3410 Boehringer Ingelheim Investigational Site, Majadahonda-Madrid
  - 1220.48.3403 Boehringer Ingelheim Investigational Site, Seville
  - 1220.48.3401 Boehringer Ingelheim Investigational Site, Valencia
- 1220.48.4106 Boehringer Ingelheim Investigational Site, Bern, Switzerland
- 1220.48.8802 China Medical University Hospital, Taichung, Taiwan
- United Kingdom (7):
  - 1220.48.4405 Boehringer Ingelheim Investigational Site, Bristol
  - 1220.48.4409 Boehringer Ingelheim Investigational Site, London
  - 1220.48.4401 Boehringer Ingelheim Investigational Site, Manchester
  - 1220.48.4408 Boehringer Ingelheim Investigational Site, Nottingham
  - 1220.48.4407 Boehringer Ingelheim Investigational Site, Oxford
  - 1220.48.4403 Boehringer Ingelheim Investigational Site, Southampton
  - 1220.48.4404 Boehringer Ingelheim Investigational Site, Tooting, London

REFERENCES:
- [Derived] Foster GR, Ferenci P, Asselah T, Mantry P, Dufour JF, Bourliere M, Forton D, Maevskaya M, Wright D, Yoshida EM, Garcia-Samaniego J, Oliveira C, Wright M, Warner N, Sha N, Quinson AM, Stern JO. Open-label study of faldaprevir plus peginterferon and ribavirin in hepatitis C virus genotype 1-infected patients who failed placebo plus peginterferon and ribavirin. J Viral Hepat. 2016 Mar;23(3):227-31. doi: 10.1111/jvh.12485. Epub 2015 Nov 17. PMID 26572686

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-national, open-label trial enrolling two cohorts of patients with chronic Hepatitis C Virus (HCV) infection of genotype 1 (GT-1) who were randomized to the placebo arm (+ Pegylated interferon α-2a/ Ribavirin) and experienced virologic failure in one of the 1220.7 (NCT01358864), 1220.30 (NCT01343888), 1220.47 (NCT01297270) trials.
Pre-assignment Details: Eligible patients who entered the rollover trial within 14 weeks of their last study visit in one of the predecessor trials were not required to do a screening visit (treatment start: Day 1). Eligible patients who were outside of this 14-week window were required to do a screening visit (Visit 1) and started treatment at Visit 2 (Day 1).
Groups:
- Relapse: Faldaprevir (FDV) 240 mg once daily combined with Pegylated interferon α-2a (PegIFN)/ Ribavirin (RBV) for 24 weeks was administered for relapser patients.
  At week 24, patients who did not achieve early treatment success (ETS) continue with an additional 24 weeks of PegIFN/RBV.
  ETS is defined as Hepatitis C virus(HCV) Ribonucleic Acid (RNA) <25 Internalional Units (IU)/millilitre (ml) (detected or undetected) at week 4 and <25 IU/ml (undetected) at week 8.
  Patients who had undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) levels at the end of treatment in one of the previous studies (see recruitment details) but had detectable levels in subsequent assessments are called relapser.
- Non-relapse: Faldaprevir (FDV) 240mg once daily combined with Pegylated interferon α-2a (PegIFN)/ Ribavirin (RBV) for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV for non-relapser patients.
  Non-relapser are non-responder (null and partial) and breakthrough patients. Null responders are patients who did not achieve > 2 log10 decrease in HCV RNA from baseline during the treatment period.
  Partial non-responders are patients who achieved > 2 log10 decrease in HCV RNA from baseline but who never achieved an undetectable level of HCV RNA.
  Breakthrough are patients who achieved an undetectable HCV RNA during the treatment period but had detectable HCV RNA at the end of treatment.
Period: Overall Study
Arm/Group | Relapse | Non-relapse
Started | 43 | 75
Completed | 41 | 60
Not Completed | 2 | 15
Not completed — Adverse Event | 2 | 2
Not completed — Lack of Efficacy | 0 | 10
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — other than above | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): This set included all patients who entered the trial, were dispensed study medication, and were documented to have taken at least one dose of study medication.
Groups:
- Relapse: FDV 240 mg once daily combined with PegIFN/RBV for 24 weeks. At week 24, if the patients did not achieve ETS the patients received an additional 24 weeks of PegIFN/RBV.
- Non-relapse: FDV 240mg once daily combined with PegIFN/RBV for 24 weeks, followed by an additional 24 weeks of PegIFN/RBV.
- Total: Total of all reporting groups
Arm/Group | Relapse | Non-relapse | Total
Number analyzed (Participants) | 43 | 75 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (7.38) | 53.4 (9.46) | 54.1 (8.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 25 | 41
  Male | 27 | 50 | 77

OUTCOME MEASURES:

1. Primary Outcome: Sustained Virological Response (SVR): Plasma HCV RNA Level < 25 IU/mL
Description: The primary endpoint was SVR12, defined as a plasma Hepatitis C virus (HCV) Ribonucleic acid (RNA) level <25 IU/mL (undetected) 12 weeks after the originally planned treatment duration.
Time Frame: 12 weeks post treatment, up to 60 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants | 95.3 [89.1 to 100] | 54.7 [43.4 to 65.9]

2. Secondary Outcome: Sustained Virological Response After 24 Weeks of Treatment Discontinuation (SVR24)
Description: Sustained virologic response 24 weeks, defined as a plasma HCV RNA level < 25 IU/mL (undetected) 24 weeks after the originally planned treatment duration.
Time Frame: 24 weeks post treatment, up to 72 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants | 95.3 [89.1 to 100.0] | 54.7 [43.4 to 65.9]

3. Secondary Outcome: Early Treatment Success (ETS)
Description: ETS, defined as a plasma HCV RNA level <25 IU/mL (detected or undetected) at week 4 and HCV RNA <25 IU/mL (undetected) at week 8.
Time Frame: week 4 and week 8
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants | 97.7 | 65.3

4. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at End of Treatment (EoT)
Description: This will be presented as the number of patients in/not in normal range from baseline EoT. SVR12 is sustained virological response 12 weeks post-treatment.
Time Frame: Week 24 for relapsers with ETS; Week 48 for relapsers without ETS, and non-relapsers
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
participants
  SVR12 = Yes | 41 | 41
  SVR12 = Yes, Baseline Normal to EOT Normal | 12 | 10
  SVR12 = Yes, Baseline Elevated to EOT Normal | 16 | 15
  SVR12 = No | 2 | 34
  SVR12 = No, Baseline Normal to EOT Normal | 0 | 11
  SVR12 = No, Baseline Elevated to EOT Normal | 2 | 9

5. Secondary Outcome: Alanine Aminotransferase (ALT) Normalisation: ALT in Normal Range at 12 Weeks Post-treatment.
Description: This will be presented as the number of patients in/not in normal range from baseline to 12 weeks post treatment. SVR12 is sustained virological response 12 weeks post-treatment.
Time Frame: 48 weeks for relapsers with ETS; 60 weeks for non-relapsers and relapsers without ETS
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
participants
  SVR12 = Yes | 41 | 41
  SVR12 = Yes, Baseline Normal to SVR12 Normal | 12 | 11
  SVR12 = Yes, Baseline Elevated to SVR12 Normal | 27 | 27
  SVR12 = No | 2 | 34
  SVR12 = No, Baseline Normal to SVR12 Normal | 0 | 8
  SVR12 = No, Baseline Elevated to SVR12 Normal | 1 | 2

6. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at End of Treatment (EoT)
Description: This will be presented as the number of patients in/not in normal range from baseline to EoT. SVR12 is sustained virological response 12 weeks post-treatment.
Time Frame: Week 24 for relapsers with ETS; Week 48 for relapsers without ETS, and non-relapsers.
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
participants
  SVR12 = Yes | 41 | 41
  SVR12 = Yes, Baseline Normal to EOT Normal | 15 | 13
  SVR12 = Yes, Baseline Elevated to EOT Normal | 14 | 11
  SVR12 = No | 2 | 34
  SVR12 = No, Baseline Normal to EOT Normal | 1 | 12
  SVR12 = No, Baseline Elevated to EOT Normal | 1 | 7

7. Secondary Outcome: Aspartate Aminotransferase (AST) Normalisation: AST in Normal Range at 12 Weeks Post-treatment.
Description: as for outcome 5
Time Frame: Week 48 for relapsers with ETS; Week 48 for relapsers without ETS, and non-relapsers
Population: FAS
Measure: Number; unit: participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
participants
  SVR12 = Yes | 41 | 41
  SVR12 = Yes, Baseline Normal to SVR12 Normal | 15 | 14
  SVR12 = Yes, Baseline Elevated to SVR12 Normal | 22 | 24
  SVR12 = No | 2 | 34
  SVR12 = No, Baseline Normal to SVR12 Normal | 1 | 10
  SVR12 = No, Baseline Elevated to SVR12 Normal | 0 | 3

8. Secondary Outcome: Occurrence of Adverse Events (Overall and by DAIDS Grade)
Description: This outcome measure will be presented as the percentage of subjects with any adverse event (AE).
  Percentages are calculated using total number of subjects per treatment cohort as the denominator.
  The intensity of all AEs was evaluated according to the DAIDS (Division of Acquired Immunodeficiency Syndrome) grading scale with AEs of mild, moderate, or severe intensity receiving Grades 1, 2, or 3, respectively. Adverse events judged potentially life threatening received a Grade 4 assessment.
Time Frame: from first intake of study medication until 30 days after discontinuing faldaprevir, up to a maximum of 213 days
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants
  Overall | 90.7 | 93.3
  Subjects with DAIDS Grade 2, 3 or 4 AEs | 65.1 | 56.0
  Subjects with DAIDS Grade 3 or 4 AEs | 27.9 | 17.3
  Subjects with DAIDS Grade 4 AEs | 7.0 | 1.3

9. Secondary Outcome: Occurrence of Adverse Events Leading to Treatment Discontinuation
Description: This outcome measure will be presented as the percentage of subjects with adverse events leading to discontinuation of Faldaprevir and all study medication. Percentages are calculated using total number of subjects per treatment cohort as the denominator.
Time Frame: from first intake of study medication until 30 days after discontinuing faldaprevir, up to a maximum of 213 days
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants
  discontinuation of faldaprevir | 4.7 | 2.7
  discontinuation of all study medication | 2.3 | 0.0

10. Secondary Outcome: Occurrence of Serious Adverse Events (SAEs)
Description: This outcome measure will be presented as the percentage of subjects with any serious adverse event (SAE). Percentages are calculated using total number of subjects per treatment cohort as the denominator.
Time Frame: from first intake of study medication until 30 days after discontinuing faldaprevir, up to a maximum of 213 days
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants | 2.3 | 8.0

11. Secondary Outcome: Occurrence of Drug-related AEs as Assessed by the Investigator
Description: This outcome measure will be presented as the percentage of subjects with any drug-related AEs as assessed by the investigator. Percentages are calculated using total number of subjects per treatment cohort as the denominator.
Time Frame: from first intake of study medication until 30 days after discontinuing faldaprevir, up to a maximum of 213 days
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants | 88.4 | 88.0

12. Secondary Outcome: Laboratory Test Abnormalities by DAIDS Grades
Description: This Outcome measure will be presented as summary of the percentage of patients with worst on-treatment Division of Acquired Immunodeficiency Syndrome (DAIDS) grade laboratory abnormalities for selected analytes (Haemoglobin, Alanine aminotransaminase (ALT), Aspartate aminotransaminase (AST) and Bilirubin total) with particular relevance to patients with HCV.
Time Frame: baseline (day 1, after first dose of randomised treatment) up to 7 days after the last intake of study
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
percentage of participants
  Haemoglobin, Grade 2 | 14.0 | 18.9
  Haemoglobin, Grade 3 | 11.6 | 8.1
  Haemoglobin, Grade 4 | 0.0 | 0.0
  ALT, Grade 2 | 7.0 | 6.7
  ALT, Grade 3 | 2.3 | 4.0
  ALT, Grade 4 | 2.3 | 0.0
  AST, Grade 2 | 4.7 | 10.7
  AST, Grade 3 | 2.3 | 2.7
  AST, Grade 4 | 2.3 | 0.0
  Bilirubin, total, Grade 2 | 32.6 | 37.3
  Bilirubin, total, Grade 3 | 39.5 | 29.3
  Bilirubin, total, Grade 4 | 11.6 | 13.3

13. Secondary Outcome: Changes From Baseline in Laboratory Test Values Over Time [Haemoglobin]
Description: This outcome measure will be presented as the mean value and the standard deviation at baseline, week 4, week 12, the minimum (min) value on treatment, maximum (max) value on treatment and last measured value on treatment. Analytes with particular relevance for patients with HCF have been selected: Haemoglobin, Alanine aminotransaminase (ALT), Aspartate aminotransaminase (AST) and Bilirubin total.
  In this outcome measure Haemoglobin is presented.
Time Frame: baseline (the last observed measurement prior to administration of any randomised study medication), week 4, week 12 (after start of treatment)
Population: FAS
Measure: Mean (Standard Deviation); unit: gram (g)/decilitre (dL)
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
gram (g)/decilitre (dL)
  Baseline (N=43, 74) | 14.8 (1.3) | 14.8 (1.4)
  week 4 (N=41, 69) | 12.6 (1.6) | 12.7 (1.4)
  week 12 (N=43, 66) | 11.7 (1.6) | 11.5 (1.5)
  min value on treatment (N=43, 74) | 11.1 (1.5) | 11.3 (1.7)
  max value on treatment (N=43, 74) | 13.7 (1.2) | 14.0 (1.4)
  last value on treatment (N=43, 74) | 11.4 (1.5) | 11.8 (1.6)

14. Secondary Outcome: Changes From Baseline in Laboratory Test Values Over Time [ALT]
Description: This outcome measure will be presented as the mean value and the standard deviation at baseline, week 4, week 12, the minimum (min) value on treatment, maximum (max) value on treatment and last measured value on treatment. Analytes with particular relevance for patients with HCF have been selected: Haemoglobin, Alanine aminotransaminase (ALT), Aspartate aminotransaminase (AST) and Bilirubin total.
  In this outcome measure ALT is presented.
Time Frame: as for outcome 13
Population: FAS
Measure: Mean (Standard Deviation); unit: Units (U)/Litre (L)
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
Units (U)/Litre (L)
  Baseline (N=43, 75) | 72 (79) | 88 (63)
  week 4 (N=43, 73) | 51 (71) | 57 (49)
  week 12 (N=43, 67) | 43 (40) | 55 (62)
  min value on treatment (N=43, 75) | 30 (20) | 39 (38)
  max value on treatment (N=43, 75) | 68 (91) | 70 (62)
  last value on treatment (N=43, 75) | 40 (26) | 54 (52)

15. Secondary Outcome: Changes From Baseline in Laboratory Test Values Over Time [AST]
Description: This outcome measure will be presented as the mean value and the standard deviation at baseline, week 4, week 12, the minimum (min) value on treatment, maximum (max) value on treatment and last measured value on treatment. Analytes with particular relevance for patients with HCF have been selected: Haemoglobin, Alanine aminotransaminase (ALT), Aspartate aminotransaminase (AST) and Bilirubin total.
  In this outcome measure AST is presented.
Time Frame: as for outcome 13
Population: FAS
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
U/L
  Baseline (N=43, 75) | 54 (41) | 68 (42)
  week 4 (N=43, 73) | 48 (71) | 46 (33)
  week 12 (N=43, 67) | 41 (37) | 48 (45)
  min value on treatment (N=43, 75) | 30 (16) | 35 (25)
  max value on treatment (N=43, 75) | 63 (89) | 62 (50)
  last value on treatment (N=43, 75) | 40 (23) | 49 (39)

16. Secondary Outcome: Changes From Baseline in Laboratory Test Values Over Time [Bilirubin Total]
Description: This outcome measure will be presented as the mean value and the standard deviation at baseline, week 4, week 12, the minimum (min) value on treatment, maximum (max) value on treatment and last measured value on treatment. Analytes with particular relevance for patients with HCF have been selected: Haemoglobin, Alanine aminotransaminase (ALT), Aspartate aminotransaminase (AST) and Bilirubin total.
  In this outcome measure Bilirubin total is presented.
Time Frame: as for outcome 13
Population: FAS
Measure: Mean (Standard Deviation); unit: milligram (mg)/dL
Arm/Group | Relapse | Non-relapse
Number analyzed (Participants) | 43 | 75
milligram (mg)/dL
  Baseline (N=43, 75) | 0.5 (0.2) | 0.5 (0.2)
  week 4 (N=43, 74) | 2.8 (1.6) | 2.6 (1.7)
  week 12 (N=43, 67) | 2.7 (1.8) | 2.7 (1.9)
  min value on treatment (N=43, 75) | 1.9 (1.3) | 1.9 (1.5)
  max value on treatment (N=43, 75) | 3.6 (2.1) | 3.5 (2.2)
  last value on treatment (N=43, 75) | 2.6 (1.8) | 2.6 (1.9)

ADVERSE EVENTS:
Time Frame: from first intake of study medication until 30 days after discontinuing faldaprevir, up to a maximum of 213 days
Arm/Group | Relapse | Non-relapse
Serious Adverse Events (participants affected / at risk) | 1/43 | 6/75
Other Adverse Events (participants affected / at risk) | 38/43 | 68/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relapse (N=43) | Non-relapse (N=75)
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Oral fungal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Relapse (N=43) | Non-relapse (N=75)
Anaemia (Blood and lymphatic system disorders) | 9 | 20
Neutropenia (Blood and lymphatic system disorders) | 2 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5
Dry eye (Eye disorders) | 1 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 8
Diarrhoea (Gastrointestinal disorders) | 14 | 21
Dry mouth (Gastrointestinal disorders) | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 22 | 34
Stomatitis (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 11 | 15
Asthenia (General disorders) | 7 | 13
Chills (General disorders) | 3 | 2
Fatigue (General disorders) | 14 | 11
Influenza like illness (General disorders) | 5 | 4
Malaise (General disorders) | 1 | 6
Pyrexia (General disorders) | 4 | 8
Hyperbilirubinaemia (Hepatobiliary disorders) | 12 | 6
Jaundice (Hepatobiliary disorders) | 5 | 10
Urinary tract infection (Infections and infestations) | 3 | 1
Haemoglobin decreased (Investigations) | 3 | 1
Weight decreased (Investigations) | 3 | 3
Decreased appetite (Metabolism and nutrition disorders) | 3 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 9
Dizziness (Nervous system disorders) | 3 | 5
Dysgeusia (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 10 | 15
Depression (Psychiatric disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 5 | 14
Irritability (Psychiatric disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 8
Eczema (Skin and subcutaneous tissue disorders) | 1 | 5
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 23
Rash (Skin and subcutaneous tissue disorders) | 12 | 21
Hypertension (Vascular disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.